CLINICAL TRIAL: NCT06920810
Title: Efficacy and Safety of Viscum Album in Patients With Triple-negative Breast Cancer Undergoing Immune Checkpoint Inhibitors
Brief Title: Viscum Album for TNBC on Adjuvant Pembrolizumab
Acronym: TNBNOBA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ilsan Cha hospital (Other)
Responsible Party: Principal Investigator, Myung Han Hyun, Assistant professor, Ilsan Cha hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICICC-CT-24-02
Record Dates: First submitted 2025-03-27; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: triple negative breast cancer; adjuvant chemotherapy; pembrolizumab; mistletoe
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: viscum album group added on adjuvant pembrolizumab and adjuvant pembrolizumab monotherapy group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Viscum album group (Experimental): Viscum album Active Ingredient: Viscum album Formulation: a colorless ampoule; the solution is colorless to pale yellow and clear.
  Manufacturer: LB Abnoba Co., Ltd. Dosage and Administration: Administered subcutaneously three times per week, with dose escalation
  Interventions: Drug: viscum album
- Wait-list control group (No Intervention): Participants assigned to the waitlist control group will receive pembrolizumab monotherapy as part of their standard adjuvant chemotherapy regimen without additional investigational intervention for the first 18 weeks of the study. On week 19, Participants will begin Viscum album administration for four weeks, as the same schedule with the Viscum album group.

INTERVENTIONS:
Drug: viscum album — Active Ingredient: Viscum album Excipients: Ascorbic acid, disodium phosphate dihydrate, monosodium phosphate monohydrate Formulation: Injectable solution contained in a colorless ampoule; the solution is colorless to pale yellow and clear.
  Manufacturer: LB Abnoba Co., Ltd. Dosage and Administration: Administered subcutaneously three times per week, with dose escalation according to the following protocol.
  Arms: Viscum album group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Viscum album extract when used in combination with pembrolizumab as adjuvant chemotherapy in adult patients (aged 19 and older) who have been diagnosed with malignant neoplasm of unilateral breast and have completed surgery.

The main questions it aims to answer are:

Does the addition of Viscum album improve clinical outcomes when combined with pembrolizumab as adjuvant chemotherapy? Is Viscum album safe and tolerable for use in this patient population?

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the efficacy and safety of Viscum album extract when used in combination with pembrolizumab as adjuvant chemotherapy in adult patients (aged 19 and older) who have been diagnosed with malignant neoplasm of unilateral breast and have completed surgery.

This clinical trial aims to recruit 40 adult participants aged 19 years or older who have been diagnosed with malignant neoplasm of the unilateral breast and require adjuvant chemotherapy, including immune checkpoint inhibitors, after completing surgical tumor resection and radiotherapy.

Potential participants will receive a full explanation of the study's purpose and procedures and will voluntarily provide written informed consent. After screening for eligibility based on inclusion and exclusion criteria, only those who meet the criteria will be enrolled and proceed with the study.

Participants in the treatment group will receive Viscum album concurrently with pembrolizumab as part of their adjuvant chemotherapy regimen for 18 weeks in order to evaluate the efficacy and safety of Viscum album. Participants in the waitlist control group will undergo scheduled assessments without any additional intervention for the first 18 weeks, followed by a 4-week intervention phase starting from week 19.

Researchers will compare the treatment group receiving pembrolizumab plus 18 weeks of Viscum album to the waitlist control group, who will not receive any intervention for the first 18 weeks, to see if early administration of Viscum album leads to better outcomes compared to delayed intervention.

Participants will:

Sign informed consent after receiving full explanation of the study Be screened for eligibility based on inclusion and exclusion criteria If eligible, participants will be assigned to either the treatment or control group Receive subcutaneous injections of Viscum album three times per week for 18 weeks (treatment group only) Undergo scheduled clinical assessments throughout the study period

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older
2. Histologically confirmed diagnosis of triple-negative breast cancer
3. ECOG Performance Status of 0 or 1
4. Completed surgery and radiotherapy for localized disease, and either (a) requires adjuvant chemotherapy including immune checkpoint inhibitors, or (b) has initiated such therapy within 3 cycles
5. Laboratory values meeting the following criteria:

   Absolute Neutrophil Count (ANC) ≥ 1,500/μL Platelet count (PLT) ≥ 100,000/μL Hemoglobin (Hb) ≥ 9.0 g/dL Albumin ≥ 3.0 g/dL Acceptable levels of creatinine, total bilirubin, AST, and ALT ≤ 3 × upper limit of normal (ULN)
6. Able to understand the study information and voluntarily provide written informed consent

Exclusion Criteria:

1. Presence of distant metastasis
2. Uncontrolled pleural effusion, ascites, or pericardial effusion
3. Other non-cancer comorbidities (e.g., dementia, cerebrovascular disease, end-stage renal disease) that are expected to significantly impair physical function
4. Pregnant or breastfeeding women
5. Estimated life expectancy of less than 3 months, making adequate follow-up unlikely
6. Any other medical condition that may interfere with study results or any situation in which, in the investigator's judgment, participation is not appropriate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
cytokine panel | week 1, week 4, week 7, week 19
  the result of immune-related cytokine panel kit (CCL2, CCL3, CCL4, CD40 Ligand, CXCL10, GM-CSF, Granzyme B, IFN-α, IFN-γ, IL-1α, IL-1β, IL-1ra, IL-2, IL-4, IL-6, IL-8, IL-9, IL-10, IL-12 p70, IL-13, IL-15, IL-17, IL-33, PD-L1, TNF-α)

SECONDARY OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 | week 1, week 4, week 7, week 19
  The EORTC QLQ-C30 is a validated, widely used questionnaire developed by the European Organisation for Research and Treatment of Cancer to assess health-related quality of life in cancer patients. It includes 30 items covering functional status, symptoms, and global health and has been validated across multiple languages and cancer populations.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Breast 23 | week 1, week 4, week 7, week 19
  The EORTC QLQ-BR23 is a validated breast cancer-specific module designed to be used alongside the EORTC QLQ-C30. It includes 23 items that assess breast cancer-related symptoms, treatment side effects, body image, and sexual functioning, and has been validated in diverse cultural and clinical settings.
MD Anderson Symptom Inventory - core | week 1, week 4, week 7, week 19
  The MD Anderson Symptom Inventory (MDASI) is a validated patient-reported outcome measure developed by MD Anderson Cancer Center to assess the severity of cancer-related symptoms and their impact on daily functioning. It consists of 13 symptom severity items and 6 interference items.

CONTACTS AND LOCATIONS:
Locations (1):
- Ilsan Cha Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data due to institutional policy and/or the sensitive nature of the clinical data collected. Future sharing may be considered on a case-by-case basis pending appropriate approvals.